CLINICAL TRIAL: NCT05854797
Title: Comparison of Normal Walking Vs Brisk Walking on Body Fat, Hypertension, Diabetes, and Level of Happiness in Over-Weight Adults.
Brief Title: Comparison Of Normal Walking Vs Brisk Walking In Over-Weight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01412 SADIA MUNAWAR
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Overweight; Walking
Keywords: Blood Pressure; Blood Glucose; Walking; Body Mass Index; Physical Activity; Exercise
MeSH Terms: conditions — Overweight; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Walking Group (Active Comparator): Adhering to FITT method, normal walking will be performed 5 days a week (frequency) to ensure optimal results. Speed (intensity) for normal will be 3.5 mph
  Interventions: Other: Normal Walking
- Brisk Walking Group (Experimental): Adhering to FITT method, brisk walking will be performed 5 days a week (frequency) to ensure optimal results. Speed (intensity) for normal will be 4.5 mph.
  Interventions: Other: Brisk Walking

INTERVENTIONS:
Other: Normal Walking — Adhering to FITT method, normal walking will be performed 5 days a week (frequency) to ensure optimal results. Speed (intensity) for normal will be 3.5 mph. The pulse rate of participants will be monitored through treadmill monitor. The duration (time) of walk each day will be 30 minutes.
  Measurement of body fat percentage, hypertension, diabetes, and level of happiness (at the beginning and ending of twelve weeks)
  Arms: Normal Walking Group
Other: Brisk Walking — Adhering to FITT method, brisk walking will be performed 5 days a week (frequency) to ensure optimal results. Speed (intensity) for normal will be 4.5 mph. The pulse rate of participants will be monitored through treadmill monitor. The duration (time) of walk each day will be 30 minutes.
  Measurement of body fat percentage, hypertension, diabetes, and level of happiness (at the beginning and ending of twelve weeks)
  Arms: Brisk Walking Group

SUMMARY:
The goal of this clinical trial is to see the comparison of normal walking vs brisk walking on body fat, hypertension, diabetes, and level of happiness in over-weight adults. The main question it aims to answer is:

Will there be a difference between the effectiveness of normal walking and brisk walking on improving body fat, hypertension, diabetes, and level of happiness in over-weight adults..

The participants will be divided into two groups; group A and group B. Group A will perform normal walk and Group B will perform brisk walk.

DETAILED DESCRIPTION:
In the modern times, despite the fact that the benefits of regular physical activity are widely known, the choice of a sedentary lifestyle is increasing in prevalence. With the help of simple and natural movements, walking is considered as a moderate level of workout intensity that promotes a long and healthy lifespan. Meanwhile, it provides the added advantage to individuals by reducing chances of injury, making it an excellent choice for middle-aged and elderly individuals. Walking tends to be the widely preferred choice of most diabetic patients worldwide for improving glycemic control. Moghetti et al. showed the correlation between walking and type 2 diabetes in their recent research where they employed meta-analysis (supported with short and long term RCTs) to prove that sufficient amount of walking can lead to improved levels of HbA1c. Walking can improve functional capacity of people with T2DM and cast favorable impacts on chronic complications of diabetes The research carried out to advocate strong relation between walking and healthy lifestyle is widely available to us. However, it mainly focuses on elderly people (with age above 60) instead of young and middle-aged people who have been equally pushed at the verge of risks to develop obesity, cardiovascular diseases and T2D due to astonishingly common sedentary lifestyle prevailing in today's world. Also, it is limited in terms of defined intensities for walking and their comparison for guiding an appropriate course of action for obese or hypertensive adults. Therefore, this research will evaluate and compare the impacts of normal and brisk walking on middle-aged people struggling with diabetes, hypertension, obesity or other cardiovascular diseases. Also, it will define the basis for a well-informed and focussed approach to enhance quality of life in adults.

ELIGIBILITY:
Inclusion Criteria:

* Age between 36-55 years
* Hypertensive middle-aged adults
* BMI > 25
* Type 2 diabetes middle-adults
* Body fat > 25%

Exclusion Criteria:

* Severe psychological illness
* Physical defect or deformity
* Experience of diabetic coma
* Engagement in other training programs
* Any other serious illness like TB, cancer.

Ages: 36 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Body Fat | 12 Weeks
  Skin fold caliper will be used for measuring body fat having reliability index of 96%. Validations of these results are costly using dual-energy x-ray absorptiometry (DXA) or hydrostatic weighing. Therefore, pre-published articles shall be taken as basis for employment of skin fold calipers to measure body fat.
Blood Pressure | 12 Weeks
  A properly calibrated sphygmomanometer with initial mercury reading at 0 will be used for measuring blood pressure. The reliability of sphygmomanometer is measured at 83% with only 4% showing a difference of more than 10 mm Hg. Both manual and digital sphygmomanometer shall be used to validate the final result.
Blood Glucose | 12 Weeks
  Red blood cells live for up to 3 months, so HbA1c gives an indication of how much sugar there has been in the blood over the past few months. It's different to the blood glucose test, which measures how much sugar is in the blood at that moment. The sensitivity and specificity ranged from 24% to 78% and 79% to 100% respectively for HbA1c (6.5%) for diagnosis of diabetes.
Level of Happiness | 12 Weeks
  Oxford happiness questionnaire has been a widely adopted tool for measuring quality of life and happiness index. The assessed reliability by test-retest after 3 weeks using Oxford happiness questionnaire has been 79% .
Body Mass Index | 12 Weeks
  Body Mass Index is a reliable indicator of body fat based on height and weight of an adult. These BMI values can be calculated free by using online calculators available at NHS (UK) and NHLBI (USA).

CONTACTS AND LOCATIONS:
Overall Officials: Jawad Naweed, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Polymed, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No